CLINICAL TRIAL: NCT00210145
Title: Impact of a Socio-aesthetic Intervention on Body Image and Quality of Life in Patients With Mastectomy or Tumorectomy for Breast Cancer.
Brief Title: Socio-aesthetic Intervention on Body Image and Quality of Life in Women With Breast Cancer.
Acronym: ASE K SEIN
Status: Withdrawn | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2003-22; ASE K SEIN
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Aesthetic care,; Mastectomy,; Breast cancer,; Quality of life,; Body image,; Psychological adjustment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Aesthetic care

SUMMARY:
The aim of this study is to evaluate the impact of a socio-aesthetic intervention on body image and quality of life in post-surgical patients with mastectomy or tumorectomy for breast cancer.Two groups of randomized subjects were constituted. Patients of the experimental group received 2 or 3 aesthetic care during the first post-surgical week, whereas those of the control group not. Body image, quality of life and diverse other personality variables were assessed at three different times: surgical operation day before, exit day before of hospitalization and three months afterwards. Our general hypothesis is that subjects who receive aesthetic care report levels significantly higher of corporal satisfaction and of quality of life at the end of the hospitalization and three months later than patients of the control group.

ELIGIBILITY:
Inclusion criteria:

First diagnosis of cancer and first surgical treatment for cancer Diagnosis of breast cancer

Exclusion criteria:

Psychiatric antecedents Inclusion in another psychosocial research

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-10 (Actual); Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice LAKDJA, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No